CLINICAL TRIAL: NCT04907045
Title: Digital Therapeutics for Opioids and Other Substance Use Disorders in Primary Care Pilot (DIGITS Trial Pilot)
Brief Title: An Initial Study of the Implementation of Digital Therapeutics for Substance Use Disorders in Primary Care
Acronym: DIGITS Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 218046; R01DA047954 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Drug Use Disorders; Illicit Drug Use; Alcohol-Related Disorders
Keywords: Implementation Science; Mobile Applications; Drug Use Disorders; Quality Improvement; Primary Health Care
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders

STUDY DESIGN:
Intervention Model Description: Non-randomized parallel groups pilot study to evaluate intervention delivery, data collection, and analysis procedures. Two primary care clinics will implement the reSET and reSET-O digital therapeutics for substance use disorders. There will be one clinic per arm in this pilot study. Implementation strategies will be varied across arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Implementation Plus Health Coaching (Experimental): The clinic in this arm will implement reSET and reSET-O with a standard implementation strategy and patients at the clinic will receive support from a health coach to help them engage with reSET and reSET-O.
  Interventions: Behavioral: Health Coaching; Behavioral: Standard Implementation
- Standard Implementation Plus Health Coaching and Practice Facilitation (Experimental): The clinic in this arm will implement reSET and reSET-O with a standard implementation strategy and patients at the clinic will receive support from a health coach to help them engage with reSET and reSET-O. Additionally, a practice facilitator will provide the clinic with support for implementation.
  Interventions: Behavioral: Health Coaching; Behavioral: Practice Facilitation; Behavioral: Standard Implementation

INTERVENTIONS:
Behavioral: Health Coaching — The clinic is provided access to a health coach who conducts outreach with patients. The health coach facilitates engagement with the digital therapeutic and encourages contact with the care team.
Behavioral: Practice Facilitation — In the context of a supportive relationship, a trained facilitator delivers the following interventions to clinic staff: Bolster Education, Audit and Provide Feedback, Support Plan-Do-Study-Act Cycles, Engage Others in Change.
  Arms: Standard Implementation Plus Health Coaching and Practice Facilitation
Behavioral: Standard Implementation — Brief clinician training and an implementation toolkit consisting of job aids, patient educational materials, scripted conversations, electronic health record tools, and a population management workbench.

SUMMARY:
The DIGITS Trial addresses a critical knowledge gap: How to best implement digital treatments for opioids and other substance use disorders in primary care. In this pilot study, the FDA-authorized reSET and reSET-O digital therapeutics will be implemented in 2 primary care clinics as part of quality improvement. The pilot is comprised of a 3-month period in which a standard approach to implementing reSET and reSET-O is applied in the two primary care clinics "standard implementation", followed by a second 3-month period in which the study will test and refine the two experimental implementation strategy interventions, health coaching (patient-facing) and practice coaching (clinician-facing) in the same clinics. This study will also pilot economic data collection tools and collect qualitative data for a formative evaluation. The analytic goals are to inform the statistical design and data collection processes for the subsequent cluster-randomized DIGITS Trial.

ELIGIBILITY:
Inclusion Criteria:

* Had a primary care visit in a participating clinic during the pilot
* Screened positive for substance use
* Adult aged 18 years or older at time of visit

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1552 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Glass, PhD, MSW, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mogk J, Idu AE, Bobb JF, Key D, Wong ES, Palazzo L, Stefanik-Guizlo K, King D, Beatty T, Dorsey CN, Caldeiro RM, Garza McWethy A, Glass JE. Prescription Digital Therapeutics for Substance Use Disorder in Primary Care: Mixed Methods Evaluation of a Pilot Implementation Study. JMIR Form Res. 2024 Sep 2;8:e59088. doi: 10.2196/59088. PMID 39222348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected from the Electronic Health Record (EHR) for an accrual period and an outcomes assessment period.
Pre-assignment Details: Of the 18,577 primary care patients with visits to the eligible clinics, 1,552 were eligible for the analysis.
Period: Overall Study
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation
Started | 296 | 1256
Prescribed (Prescribed represents the number of patients prescribed the digital therapeutic. While this is a study outcome, we have added it as a study milestone, because it represents the population for which adverse events were monitored.) | 6 | 8
Completed | 296 | 1256
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation | Total
Number analyzed (Participants) | 296 | 1256 | 1552
Age, Customized [Count of Participants; unit: Participants]
  Age group: 18-24 years | 60 | 182 | 242
  Age group: 25-34 years | 153 | 459 | 612
  Age group: 35-44 years | 48 | 218 | 266
  Age group: 45-54 years | 13 | 126 | 139
  Age group: =>55 years | 22 | 271 | 293
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 635 | 795
  Male | 136 | 621 | 757
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 89 | 114
  Not Hispanic or Latino | 163 | 899 | 1062
  Unknown or Not Reported | 108 | 268 | 376
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 25 | 67 | 92
  Race: Black or African American | 17 | 54 | 71
  Race: White | 179 | 916 | 1095
  Race: Multiple race | 19 | 54 | 73
  Race: Other race, combined to maintain patient confidentiality | 15 | 65 | 80
  Race: Missing race data | 41 | 100 | 141
Rurality of residence [Count of Participants; unit: Participants] — Rurality and urbanity was defined using the 2010 rural-urban commuting area codes and 2010 Census Tract geocoding
  Participants
    Urban | 296 | 1255 | 1551
    Rural | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Reach of the Digital Therapeutic to Patients in the Primary Care Clinic
Description: The proportion of patients who initiate the digital therapeutic, defined by instances in which patients open the app, enter the prescription code, and use a treatment module
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation
Number analyzed (Participants) | 296 | 1256
Participants | 1 | 4

2. Primary Outcome: Fidelity of Patients Use of the Digital Therapeutic to Clinical Recommendations
Description: Mean number of weeks in which patients use 4 app modules/week and have visited a clinician in the past month
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Number of weeks
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation
Number analyzed (Participants) | 296 | 1256
Number of weeks | 0 (0.06) | 0 (0.06)

3. Secondary Outcome: Effectiveness
Description: Mean number of months in which patients make monthly visits for substance use disorder
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Number of months
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation
Number analyzed (Participants) | 296 | 1256
Number of months | 0.01 (0.12) | 0 (0.06)

4. Other Pre Specified Outcome: Reach-3
Description: The proportion of patients who download and unlock reSET or reSET-O
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation
Number analyzed (Participants) | 296 | 1256
Participants | 1 | 6

5. Other Pre Specified Outcome: Reach-2
Description: The proportion of patients prescribed reSET or reSET-O
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation
Number analyzed (Participants) | 296 | 1256
Participants | 6 | 8

6. Other Pre Specified Outcome: Fidelity-2
Description: Mean number of weeks in which patients use at least 1 module/week
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Number of weeks
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation
Number analyzed (Participants) | 296 | 1256
Number of weeks | 0 (0.06) | .01 (.35)

7. Other Pre Specified Outcome: Fidelity-3
Description: Mean number of weeks in which patients use at least 4 modules/week
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Number of weeks
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation
Number analyzed (Participants) | 296 | 1256
Number of weeks | 0 (0.06) | 0 (0.06)

ADVERSE EVENTS:
Time Frame: From date of prescription through end of prescription (approximately 90 days).
Arm/Group | Standard Implementation Plus Health Coaching | Standard Implementation Plus Health Coaching and Practice Facilitation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04907045/Prot_SAP_000.pdf